CLINICAL TRIAL: NCT06408051
Title: Efficacy of 200 IU OnabotulinumtoxinA (Botulinum Toxin Type A) in Patients With Idiopathic
Brief Title: Efficacy of 200 IU OnabotulinumtoxinA in Idiopathic Overactive Bladder Resistant to Anticholinergic Treatment
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Principal Investigator, Hisar Intercontinental Hospital
Other Study IDs: 10.11.203/23-54
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Overactive Bladder Resistant to Anticholinergic Treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- singel
  Interventions: Procedure: Injection of onabotulinumtoxinA into the bladder wall

INTERVENTIONS:
Procedure: Injection of onabotulinumtoxinA into the bladder wall — BTX was injected into the detrusor muscles at 20 sites

SUMMARY:
This study aimed to assess the efficacy and safety of onabotulinumtoxinA (botulinum toxin type A) in patients with idiopathic overactive bladder (OAB) and urinary incontinence who had previously failed to respond to anticholinergic treatment. Additionally, we examined the impact of significant reductions in bladder wall thickness on therapeutic outcomes.

DETAILED DESCRIPTION:
The efficacy of OnabotulinumtoxinA was investigated in patients who attended urology outpatient clinics between January 2016 and June 2022 for overactive bladder unresponsive to anticholinergic therapy. Baseline symptoms and quality of life data were compared to those at month 6 after the treatment. The voiding diary (for 3 days) of each patient was reviewed to assess and record patients' symptoms. Baseline ultrasound (US)-measured post-void residual urine (PVR) and bladder wall thickness (BWT) values were recorded. Patients with a history of neurological disorders, anticholinergic-naive patients, patients diagnosed with bladder cancer, and those with bladder outlet obstruction were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* overactive bladder urge incontinence

Exclusion Criteria:

* neurological and/or neurosurgical disorders, anticholinergic-naive patients, bladder cancer, bladder stone, interstitial cystitis, prostate cancer chronic prostatitis bladder outlet obstruction

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In patients with overactive bladder and urinary incontinence who had previously failed to respond to anticholinergic treatments
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
frequencies of urination, nocturia, incontinence episodes | 1 years
  below 8,above 8
urgency, | 1 years
  present or absent

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Basri Cakiroglu, Istanbul
  - Hisar Intercontinental Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided